CLINICAL TRIAL: NCT02280278
Title: The Effectiveness and Safety of Adjuvant Cytokine-induced Killer Cell Immunotherapy for Stage III Colorectal Cancer Patients After Chemotherapy
Brief Title: Cytokine-induced Killer Cell Immunotherapy for Surgical Resected Stage III Colorectal Cancer Patients After Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Jun Wu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5010010
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Stage III Colon Cancer
Keywords: colon cancer; cytokine-induced killer cell immunotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIK group (Experimental): Stage III Colon Cancer patients after radical operation and adjuvant chemotherapy will receive 8 cycles of CIK therapy in this group.
  Interventions: Procedure: Radical surgery; Drug: Adjuvant chemotherapy; Biological: Cytokine-induced killer cell immunotherapy
- Control group (Active Comparator): Stage III Colon Cancer patients will only receive radical operation and adjuvant chemotherapy.
  Interventions: Procedure: Radical surgery; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Procedure: Radical surgery
Drug: Adjuvant chemotherapy
Biological: Cytokine-induced killer cell immunotherapy
  Arms: CIK group

SUMMARY:
We hypothesize through this randomized, prospective, single center adjuvant study, that cytokine-induced killer cell in patients with stage III colon cancer can improve survival in this patient population over control. Stage III colon cancer patients can benefit most from adjuvant chemotherapy, but the 5 year survival rate is still around 60%. We wish CIK cell therapy can improve the survival rate of stage III colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient of ≥ 18 years of age or ≥ country's legal age for adult consent
* Stage III colon cancer
* undergone complete resection of primary tumor
* Completed standard adjuvant chemotherapy
* within 120 days of completion of standard therapy
* ECOG performancer status 0-2
* Satisfactory haematological or biochemical functions (tests should be carried out within 8 weeks prior to randomisation): Results of clinical investigations carried out within 8 weeks prior to randomisation can be used in place of the required screening investigations. Patients with mild laboratory abnormalities can be included at the discretion by the site principal investigator, and after approval by ASCOLT Trial Management Group
* ANC ≥ 1.0 x 109/L
* Platelets ≥ 100 x 109/L
* Creatinine clearance ≥ 30 mL/min
* Total bilirubin ≤ 2.0 x the upper limit normal
* AST & ALT ≤ 5 x the upper limit normal
* Completed the following investigations
* Completed the following investigations

Exclusion Criteria:

* HIV positive or other Immunodeficiency disease
* recently use of high dose glucocorticoid
* Uncontrolled hypertension (untreated systolic blood pressure > 160 mmHg, or diastolic blood pressure > 95 mmHg)
* History of recent cancers (except for colorectal cancers, non-melanoma skin cancers, basal cell carcinomas, squamous cell carcinomas) in the past 5 years
* Patient having known allergy to capecitabine or Oxaliplatin
* Pregnant, lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
survival rate | 5 years
toxin-side effect | 1 year
  Toxin-side effect will be assessed by laboratory test, clinicians and questionary

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Wu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guagzhou, Guangdong, China